CLINICAL TRIAL: NCT06545370
Title: The Impact of Nurse-led Education on Patients With Chronic Heart Failure and Their Informal Caregivers in Optimizing the Care for Both and Improving the Clinical Outcomes of Patients
Brief Title: Nurse-led Education on Patients With Chronic Heart Failure and Their Informal Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hellenic Mediterranean University (Other)
Responsible Party: Principal Investigator, Konstantinos Giakoumidakis, Associate Professor in Clinical Nursing - Chronic Diseases Management, Hellenic Mediterranean University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 10/28.05.2024
Record Dates: First submitted 2024-07-25; First posted 2024-08-09 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: Heart failure; informal caregivers; patient outcomes; nurse-led education
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group - No Intervention Group (No Intervention): the control group (Group A) will receive standard care based on the policies and protocols of primary health care
- Intervention 1 group - Patients' education (Experimental): the first intervention group (Group B) will receive nurse-led education through oral sessions, educational materials, and regular phone calls
  Interventions: Other: Intervention 1 / Nurse-led patients' education
- Intervention 2 - Patients' and caregivers' education (Experimental): the second intervention group (Group C) will receive the described nurse-led education while caregivers also undergo training through oral sessions, phone calls, and appropriately designed educational materials
  Interventions: Other: Intervention 1 / Nurse-led patients' education; Other: Intervention 2 / Nurse-led patients' & caregivers' education

INTERVENTIONS:
Other: Intervention 1 / Nurse-led patients' education — nurse-led education through oral sessions, educational materials, and regular phone calls
  Arms: Intervention 1 group - Patients' education; Intervention 2 - Patients' and caregivers' education
Other: Intervention 2 / Nurse-led patients' & caregivers' education — nurse-led education while caregivers also undergo training through oral sessions, phone calls, and appropriately designed educational materials
  Arms: Intervention 2 - Patients' and caregivers' education

SUMMARY:
The current study intends to examine the influence of nurse-led education on patients with chronic heart failure and their caregivers, with the goal of optimizing care for both and improving patients' clinical outcomes.

DETAILED DESCRIPTION:
Introduction: Heart failure is a clinical syndrome with pandemic characteristics, and its prevalence increases with age. The development of self-care behavior by patients seems to be a crucial component for effective management and reduction of the disease's impact. Nurse- guided patient education has been associated with improved outcomes and the development of self-care behavior. In recent years, several studies have also focused on the contribution of informal caregivers to improving the outcomes of the disease. Nurse-led education for both patients and their caregivers has been shown to enhance their caregiving skills, leading to better disease management and beneficial outcomes.

Purpose: To investigate the impact of nurse-led education on patients with chronic heart failure and their caregivers, aiming to optimize care for both and improve the clinical outcomes of patients.

Methodology: A randomized controlled trial will be conducted with the manipulation of independent variables and the creation of a control group. Patients will be randomly assigned to three groups: a) the control group (Group A), receiving standard care based on the policies and protocols of primary health care; b) the first intervention group (Group B), receiving nurse-led education through oral sessions, educational materials, and regular phone calls; and c) the second intervention group (Group C), receiving the described nurse-led education while caregivers also undergo training through oral sessions, phone calls, and appropriately designed educational materials. Greek versions of the Minnesota Living with Heart Failure Questionnaire, Hippocratic Hypertension Self-Care Scale, and Self-Efficacy for Appropriate Medication Use Scale will be used to assess quality of life, self-care behavior, and medication adherence. For caregivers, their quality of life, caregiving burden, and sense of guilt will be evaluated using Greek versions of the EuroQol ED-5, Heart Failure Caregiver Questionnaire, and Caregiver Guilt Questionnaire, respectively. Measurements will be taken before patient and caregiver education (initial meeting), 1 month, and 6 months after the initial meeting. Statistical analysis will be performed using SPSS (version 26) and descriptive and inferential statistical analysis methods.

Expected Results: The proposed study is expected to highlight the contribution of nurse-led education in optimizing care for both patients and their caregivers. Additionally, this education is anticipated to lead to better clinical outcomes for patients with chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients recently hospitalized due to the disease
* Patients and caregivers who are literate in Greek
* Patients and caregivers who provide written informed consent for their participation in the study
* Patients diagnosed with heart failure for at least 6 months
* Caregivers who have been involved in the care of the patients for at least 6 months
* Patients taking medication according to the guidelines of the European Society of Cardiology

Exclusion Criteria:

* History of psychiatric disease, recent history of alcohol or/and drug abuse, dementia, and Alzheimer's disease (for patients and caregivers)
* Absence of an informal caregiver according to their statement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Heart Failure Patients' Quality of Life | from date of first communication with patient until the date of documented progression, assessed up estimate to 24 months.
  The heart failure patient's quality of life: To assess the quality of life of patients with heart failure, the Greek version of the Minnesota Living with Heart Failure Questionnaire (MLwHFQ) was used.
Heart failure patients' self-care | from date of first communication with patient until the date of documented progression, assessed up estimate to 24 months.
  The self-care behavior of heart failure patients: The Hippocratic Heart Failure Self-Care Scale is an 18-item scale created by Greek researchers (Brokalaki et al., 2024).
Medication adherence | from date of first communication with patient until the date of documented progression, assessed up estimate to 24 months.
  The adherence of pharmacological treatment to heart failure patients: To assess adherence to medication in patients with cardiac deficiency, the Greek version of SEAMS will be used (Theofilou, 2023). SEAMS is a 13-item self-report medication adherence scale.

SECONDARY OUTCOMES:
Caregivers' quality of life | From date of first communication with patient until the date of documented progression, assessed up estimate to 24 months.
  The quality of life of heart failure patients' caregivers: Assessing the quality of life of caregivers of heart failure patients will be done using the Greek version of the EuroQol EQ-5D tool (Kontodimopoulos et al., 2008).
Caregiving burden | From date of first communication with patient until the date of documented progression, assessed up estimate to 24 months.
  The burden of the heart failure patients' caregivers: The assessment of the burden of caregivers of heart failure patients will be done through the Greek version of the HF Caregiver Questionnaire.
Sense of guilt | From date of first communication with patient until the date of documented progression, assessed up estimate to 24 months.
  The sense of guilt among heart failure patients' caregivers: Assessing the guilt of caregivers of heart failure patients will be done through the Greek version of the Caregiver Guilt Questionnaire (CGQ).

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Hellenic Mediterranean University, Heraklion, Crete
  - Hellenic Mediterranean University, Heraklion

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share individual participant data (IPD) collected in this study due to concerns about patient privacy, and lack of infrastructure for data sharing